CLINICAL TRIAL: NCT05737290
Title: Effects of Clear Aligners Versus Fixed Appliances on Occlusion After Treatment of Mild Anterior Crowding: A T-scan Study.
Brief Title: Effects of Clear Aligners Versus Fixed Appliances on Occlusion After Treatment of Mild Anterior Crowding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Moaz Hafez Abdelrahman Hafez, Doctor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 893/2838
Record Dates: First submitted 2023-02-06; First posted 2023-02-21 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Occlusion
Keywords: Clear aligners; Fixed appliances; Anterior crowding; Occlusion; T scan
MeSH Terms: conditions — Bites and Stings | interventions — Orthodontic Appliances, Fixed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator)
  Interventions: Device: Clear aligners
- Group B (Active Comparator)
  Interventions: Device: Fixed appliances

INTERVENTIONS:
Device: Clear aligners — Patients with mild anterior crowding will be treated with non-extraction treatment using clear aligners.
  Arms: Group A
Device: Fixed appliances — Patients with mild anterior crowding will be treated with non-extraction treatment using fixed appliances.
  Arms: Group B

SUMMARY:
The aim of this study is to evaluate effects of clear aligners versus fixed appliances on occlusion after treatment of mild anterior crowding a T-scan study.

DETAILED DESCRIPTION:
Intervention:

Group 1. Patients treated with clear aligner. Patients with mild anterior crowding will be treated with non-extraction treatment using clear aligners.

Group 2. Patients treated with fixed appliance. Patients with mild anterior crowding will be treated with non-extraction treatment using fixed appliances.

Observations:

Multi-bite closure of left and right excursive T-Scan® recordings were obtained before and after treatment from each subject to measure the occlusal parameters to be analyzed during this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the age (14-19 y).
* Fully erupted permanent dentition, 3rd molars excluded.
* Healthy, compliant, and motivated patients who can visit the department regularly.
* Non-extraction treatment.
* Class I with mild anterior crowding lower and/ or upper.
* Good oral and general health.

Exclusion Criteria:

* Previous orthodontic treatment.
* Craniofacial abnormalities, congenital syndromes of the craniofacial area.
* Anterior or posterior crossbite.
* Anterior or lateral open bite.
* Poor oral hygiene or periodontally compromised patient.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Distribution of occlusal forces | At 6 months
  Amount of magnitude of occlusal forces after treatment by clear aligners
Distribution of occlusal forces | At 6 months
  Amount of magnitude of occlusal forces after treatment by fixed appliances

CONTACTS AND LOCATIONS:
Overall Officials: Moaz Hafez Abdelrhman, Master, Principal Investigator — Al-Azhar University
Locations (1):
- Al Azhar University, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The aim of this study is to evaluate effects of clear aligners versus fixed appliances on occlusion after treatment of mild anterior crowding a T-scan study.
Supporting Information: Study Protocol
Time Frame: 6 months

REFERENCES:
- [Background] Weir T. Invisalign treatment of lower incisor extraction cases. Aust Orthod J. 2016 May;32(1):82-7. PMID 27468595